CLINICAL TRIAL: NCT01117766
Title: A Randomized, Double Blind, Placebo Controlled, 2-Way Crossover Methodology Study Designed To Assess The Reproducibility And Sensitivity Of Quantitative Sensory Testing (QST) In Patients With Neuropathic Pain Treated With Pregabalin Vs Placebo
Brief Title: Study To Assess The Reproducibility And Sensitivity Of Quantitative Sensory Testing In Patients With Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A9011015
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2010-09-27 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Neuropathic Pain
Keywords: Methodology; Quantitative Sensory Testing; Neuropathies Pain; Pregabalin
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active drug (Active Comparator)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Dose titration according to following regimen: 75mg BID for 3 days; 150mg for 4 days; 225mg BID for 4 days; 300mg BID for 17 days. Dose reduced for renally impaired patients
  Arms: Active drug
Drug: Placebo — BID dosing for 28 days
  Arms: Placebo

SUMMARY:
Conventional pain efficacy measures such as Visual Analogue Scores (VAS) are often unable to detect treatment efficacy in small-scale clinical trials. Combining conventional pain efficacy measures with quantitative sensory testing (QST) may provide more sensitive and informative outcome measures in clinical trials.

DETAILED DESCRIPTION:
Methodology to assess reproducibility and sensitivity of quantitative sensory testing

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain of peripheral origin demonstrating spontaneous ongoing pain and dynamic mechanical allodynia to brush stimuli.
* A present pain intensity score of 4 or more (out of 10) for spontaneous ongoing pain and brush-evoked allodynia at the skin area at screen.
* Stable analgesic medication (excluding pregabalin) for a minimum of 1 month prior to the start of study.

Exclusion Criteria:

* Patients who have undergone neurolytic or neurosurgical therapy.
* Patients who have trigeminal neuralgia, central pain (due to cerebrovascular lesions, multiple sclerosis and traumatic spinal cord injuries), complex regional pain syndrome (Type I and II), and phantom limb pain.
* Patients who have previously been treated with pregabalin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Pfizer Investigational Site, Vienna, Austria
- Pfizer Investigational Site, Brussels, Belgium
- Pfizer Investigational Site, Boulogne-Billancourt, France
- United Kingdom (2):
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011015&StudyName=Study%20To%20Assess%20The%20Reproducibility%20And%20Sensitivity%20Of%20Quantitative%20Sensory%20Testing%20In%20Patients%20With%20Neuropathic%20Pain%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin Then Placebo: During the 4-week pregabalin treatment period, participants were titrated up to 300 mg twice daily (BID) for the first 2 weeks and then remained at 300 mg BID for the duration of the treatment period. Participants took a dose each morning and the evening dose approximately 12 hours later. Then after a 2-week washout period, participants took placebo to match the pregabalin doses BID during a 4-week treatment period.
- Placebo Then Pregabalin: Participants took placebo to match the pregabalin doses BID during the first 4- week treatment period. Then after a 2-week washout period, participants were titrated up to 300 mg pregabalin BID for the first 2 weeks and then remained at 300 mg BID for the duration of the second 4-week treatment period. Participants took a dose each morning and the evening dose approximately 12 hours later.
Period: First Intervention
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin
Started | 14 | 17
Received Treatment | 14 | 17
Completed | 13 | 16
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Period: Washout Period
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin
Started | 13 | 16
Completed | 13 | 14
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2
Period: Second Intervention
Arm/Group | Pregabalin Then Placebo | Placebo Then Pregabalin
Started | 13 | 14
Completed | 11 | 9
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes all participants randomized to receive pregabalin first and placebo first.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Customized [Number; unit: participants]
  18 to 44 years | 9
  45 to 64 years | 12
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Dynamic Allodynia Intensity at Visits 3 and 6 and Visits 4 and 7
Description: Five strokes applied with a standardized brush (somedic) across the painful site, 6cm long and at a control site to allow the participants to appreciate any difference. A painful and clearly dysaesthetic (unpleasant) sensation was considered as representing brush allodynia (whereas a "strange" or "tickly" sensation provoked by the brush was not). After each brush stimuli participants were asked to give a pain rating using 11-point numerical rating scale (NRS) where 0=no pain and 10=worst pain imaginable. The average of 5 brush strokes was calculated to obtain the mean score.
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: Full analysis set (FAS)=participants with present pain intensity score >=4 out of 10 for brush evoked allodynia at screening and randomization, >=4 out of 7 non missing values in week prior to randomization, >4 for weekly average daily pain score, and who did not withdraw/discontinue. n=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pregabalin: During the 4-week pregabalin treatment period, participants were titrated up to 300 mg BID for the first 2 weeks and then remained at 300 mg BID for the duration of the treatment period. Participants took a dose each morning and the evening dose approximately 12 hours later.
- Placebo: Participants took placebo to match the pregabalin doses BID.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (n=15,16) | -1.09 (1.735) | -1.16 (1.730)
  Week 4 (Visits 4 and 7) (n=18,21) | -1.31 (1.924) | -0.67 (1.984)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.7319, ANCOVA; Mean Difference (Net) = -0.19, 95% CI 2-sided [-1.29 to 0.92], Standard Error of Mean 0.537
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.3404, ANCOVA; Mean Difference (Net) = -0.52, 95% CI 2-sided [-1.61 to 0.57], Standard Error of Mean 0.536

2. Primary Outcome: Mean Change From Baseline in Dynamic Allodynia Area at Visits 3 and 6 and Visits 4 and 7
Description: Dynamic area brush in cm^2: calculated from 8 measured distances by calculating the area of an octagon. The angle between each pair of lines was 45 degrees at point c. The area of the octagon was found by totaling the areas of the 8 triangles. Octagon with 8 radial lengths from center to the outside. Area = Σ ( ½ length * perpendicular height); Σ ( ½ ri * sin(45) r(i+1) ) = Σ ( (ri * r(i+1) )/2√2)). (where ri, i=1 to 8, were the eight radial lengths)
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
cm2
  Week 3 (Visits 3 and 6) (n=16,17) | -53.441 (114.7084) | -49.180 (94.3329)
  Week 4 (Visits 4 and 7) (n=17,20) | -49.808 (100.2094) | -18.921 (104.3942)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.6539, ANCOVA; Mean Difference (Net) = -12.32, 95% CI 2-sided [-70.20 to 45.56], Standard Error of Mean 26.872
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.3678, ANCOVA; Mean Difference (Net) = -23.91, 95% CI 2-sided [-78.54 to 30.72], Standard Error of Mean 25.807

3. Primary Outcome: Mean Change From Baseline in Mechanical Pain Sensitivity (Von Frey) at Visits 3 and 6 and Visits 4 and 7
Description: Sensitivity to mechanical pain stimuli was tested using calibrated Von Frey monofilaments. To obtain a stimulus-response-function, seven different Von Frey monofilaments (size 8 to 512 mN, force increased by a factor of two from filament to filament) applied three times each; each stimulus was participant-rated using 11-point NRS where 0=no pain and 10=worst pain imaginable. If a score of 8 or more was reported for a given intensity no stronger stimuli was applied. Von Frey stimulus was applied to the skin for 1 to 2 seconds. The average of 3 ratings was calculated for the mean score.
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean. Missing values were imputed using a single imputation regression method.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (Size 8, n=15,16) | -0.133 (1.7494) | 0.417 (2.6063)
  Week 3 (Visits 3 and 6) (Size 16, n=15,16) | -1.356 (2.4800) | 0.208 (2.6412)
  Week 3 (Visits 3 and 6) (Size 32, n=15,16) | -0.200 (1.8551) | -0.188 (2.1636)
  Week 3 (Visits 3 and 6) (Size 64, n=15,16) | -1.128 (2.0304) | 0.561 (2.9543)
  Week 3 (Visits 3 and 6) (Size 128, n=15,16) | -1.267 (1.6868) | -0.097 (1.3385)
  Week 3 (Visits 3 and 6) (Size 256, n=15,16) | -0.773 (2.2420) | -0.171 (1.4133)
  Week 3 (Visits 3 and 6) (Size 512, n=15,16) | -1.533 (1.7873) | -0.480 (1.1183)
  Week 4 (Visits 4 and 7) (Size 8, n=18,21) | -0.370 (1.2674) | -0.429 (1.7132)
  Week 4 (Visits 4 and 7) (Size 16, n=18,21) | -0.611 (1.2693) | -0.889 (2.2616)
  Week 4 (Visits 4 and 7) (Size 32, n=18,21) | -0.333 (1.4597) | -0.825 (2.1386)
  Week 4 (Visits 4 and 7) (Size 64, n=18,21) | -1.116 (1.6152) | -0.462 (3.1381)
  Week 4 (Visits 4 and 7) (Size 128, n=18,21) | -1.315 (1.9322) | -0.841 (2.2843)
  Week 4 (Visits 4 and 7) (Size 256, n=18,21) | -1.322 (1.8729) | -0.751 (2.5072)
  Week 4 (Visits 4 and 7) (Size 512, n=18,21) | -1.836 (1.7249) | -0.420 (2.0238)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.0071, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = -1.09, 95% CI 2-sided [-1.84 to -0.35], Standard Error of Mean 0.342
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.1294, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = -0.59, 95% CI 2-sided [-1.36 to 0.19], Standard Error of Mean 0.370

4. Primary Outcome: Mean Change From Baseline in Punctate Allodynia Area (Von Frey) at Visits 3 and 6 and Visits 4 and 7
Description: Punctate allodynia area in cm^2: calculated from 8 measured distances by calculating the area of an octagon. The angle between each pair of lines was 45 degrees at point c. The area of the octagon was found by totaling the areas of the 8 triangles. Octagon with 8 radial lengths from center to the outside. Area = Σ ( ½ length * perpendicular height); Σ ( ½ ri * sin(45) r(i+1) ) = Σ ( (ri * r(i+1) )/2√2)). (where ri, i=1 to 8, were the eight radial lengths)
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
cm2
  Week 3 (Visits 3 and 6) (n=16,17) | -75.571 (148.8301) | -3.232 (125.8041)
  Week 4 (Visits 4 and 7) (n=17,20) | -75.834 (133.9530) | -4.130 (129.8261)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.0300, ANCOVA; Mean Difference (Net) = -61.54, 95% CI 2-sided [-116.12 to -6.96], Standard Error of Mean 25.298
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.0844, ANCOVA; Mean Difference (Net) = -49.06, 95% CI 2-sided [-105.67 to 7.55], Standard Error of Mean 26.501

5. Primary Outcome: Mean Change From Baseline in Cold Pain Sensitivity at Visits 3 and 6 and Visits 4 and 7
Description: Duration of thermal stimuli was 2 seconds and an intensity that is increased in steps of 5 degrees celsius for cold stimuli (between 5 and 20 degrees celsius). Thermal pain sensitivity was participant-rated using 11-point NRS where 0=no pain and 10=worst pain imaginable. The average of 2 ratings was calculated to get the mean score.
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (5 degrees, n=15,16) | -0.821 (1.2039) | -1.402 (3.0295)
  Week 3 (Visits 3 and 6) (10 degrees, n=15,16) | -0.333 (1.3318) | -1.313 (2.0402)
  Week 3 (Visits 3 and 6) (15 degrees, n=15,16) | -0.567 (2.3442) | 0.125 (1.3478)
  Week 3 (Visits 3 and 6) (20 degrees, n=15,16) | -0.500 (1.9365) | 0.031 (1.4314)
  Week 4 (Visits 4 and 7) (5 degrees, n=18,21) | -0.726 (1.3375) | -0.703 (2.4746)
  Week 4 (Visits 4 and 7) (10 degrees, n=18,21) | -0.278 (1.3086) | -0.810 (1.6239)
  Week 4 (Visits 4 and 7) (15 degrees, n=18,21) | -0.583 (1.2632) | 0.095 (1.5622)
  Week 4 (Visits 4 and 7) (20 degrees, n=18,21) | -0.111 (1.4507) | -0.333 (0.7130)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.7506, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.83 to 1.14], Standard Error of Mean 0.478
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.9673, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.61 to 0.64], Standard Error of Mean 0.299

6. Primary Outcome: Mean Change From Baseline in Heat Pain Sensitivity at Visits 3 and 6 and Visits 4 and 7
Description: Duration of thermal stimuli was 2 seconds and an intensity that is increased in steps of 4 degrees celsius for heat stimuli (between 40 and 50 degrees celsius). Thermal pain sensitivity was participant-rated using 11-point NRS where 0=no pain and 10=worst pain imaginable. The average of 2 ratings was calculated to get the mean score.
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (40 degrees, n=15,16) | -1.100 (2.2216) | -0.625 (2.3130)
  Week 3 (Visits 3 and 6) (44 degrees, n=15,16) | 0.400 (3.4959) | -0.938 (2.8395)
  Week 3 (Visits 3 and 6) (47 degrees, n=15,16) | -0.908 (2.5249) | -0.578 (3.3112)
  Week 3 (Visits 3 and 6) (50 degrees, n=15,16) | -1.385 (2.8981) | -0.865 (2.1050)
  Week 4 (Visits 4 and 7) (40 degrees, n=18,21) | -0.639 (2.5771) | -0.143 (0.9506)
  Week 4 (Visits 4 and 7) (44 degrees, n=18,21) | -0.444 (4.1084) | -0.495 (2.9959)
  Week 4 (Visits 4 and 7) (47 degrees, n=18,21) | -0.337 (3.0065) | -0.083 (2.7679)
  Week 4 (Visits 4 and 7) (50 degrees, n=18,21) | -0.566 (2.2423) | -0.387 (2.6689)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.5502, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.99 to 1.78], Standard Error of Mean 0.642
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.8536, ANCOVA; Statistical analysis was based on the average pain score across all levels of stimuli; Mean Difference (Net) = -0.09, 95% CI 2-sided [-1.15 to 0.96], Standard Error of Mean 0.500

7. Secondary Outcome: Mean Change From Baseline in Weekly Pain Score From the Daily Diary at Visits 3 and 6 and Visits 4 and 7
Description: Daily pain diary: participant-rated pain during the past 24 hours rated on an 11 point NRS scale where 0=no pain and 10=worst possible pain. For a given week, the pain response was the average of the 7 daily entries for that week, or average of the available data for that week if fewer than 7 entries were recorded (>=1 daily pain score for any given week required). The endpoint for each week consisted of the change from baseline in average pain score (follow-up value minus baseline).
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean. Missing weeks within a period were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (n=19,18) | -1.456 (1.8287) | -0.484 (2.0721)
  Week 4 (Visits 4 and 7) (n=18,18) | -1.397 (1.4823) | -0.769 (1.4778)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.0132, ANCOVA; Mean Difference (Net) = -1.54, 95% CI 2-sided [-2.73 to -0.34], Standard Error of Mean 0.586 — In statistical analyses, scores were further grouped to 1-3 'improved', 4 'no change' and 5-7 'worsened'
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.0403, ANCOVA; Mean Difference (Net) = -1.00, 95% CI 2-sided [-1.95 to -0.05], Standard Error of Mean 0.467 — In statistical analyses, scores were further grouped to 1-3 'improved', 4 'no change' and 5-7 'worsened'

8. Secondary Outcome: Mean Change From Baseline in Patient's Global Impression of Change (PGIC) at Visits 3 and 6 and Visits 4 and 7
Description: PGIC: participant-rated assessment measuring change in participant's overall status on a 7-point scale from 1=very much improved to 7=very much worse.
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (n=15,16) | 3.3 (1.87) | 3.4 (1.15)
  Week 4 (Visits 4 and 7) (n=18,21) | 2.4 (1.20) | 3.8 (1.63)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.6631, ANCOVA; Mean Difference (Net) = -0.19, 95% CI 2-sided [-1.12 to 0.74], Standard Error of Mean 0.433
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.0022, ANCOVA; Mean Difference (Net) = -1.54, 95% CI 2-sided [-2.48 to -0.59], Standard Error of Mean 0.465

9. Secondary Outcome: Mean Change From Baseline in Test-Day Global Pain Intensity at Visits 3 and 6 and Visits 4 and 7
Description: Global pain: participant-rated pain using the test-day global pain scale, consisting of an 11-point NRS where 0 = no pain and 10 = worst possible pain. Participants described intensity of pain in response to "How intense is your pain today?"
Time Frame: Week 3 (Visits 3 and 6) and Week 4 (Visits 4 and 7) of each period
Population: FAS. n=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale
  Week 3 (Visits 3 and 6) (n=7,10) | -1.5 (2.39) | -0.4 (2.66)
  Week 4 (Visits 4 and 7) (n=11,11) | -1.6 (1.95) | 0.0 (2.94)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 3 (Visits 3 and 6); Test type: Superiority or Other; p = 0.1753, ANCOVA; Mean Difference (Net) = -1.04, 95% CI 2-sided [-2.60 to 0.53], Standard Error of Mean 0.722
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 4 (Visits 4 and 7); Test type: Superiority or Other; p = 0.0198, ANCOVA; Mean Difference (Net) = -1.51, 95% CI 2-sided [-2.75 to -0.27], Standard Error of Mean 0.588

10. Secondary Outcome: Mean Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) Total Score at Visits 4 and 7
Description: NPSI: 10-item self-administered questionnaire assessing 5 dimensions of pain (burning superficial spontaneous pain, pressing deep spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dysesthesia). Each item consists of a question about the specific qualities of pain and an 11-point numerical scale range: 0 (absence of pain) to 10 (maximum intensity imaginable), and 2 temporal items related to spontaneous and paroxysmal pain. Maximum total score possible = 100.
Time Frame: Week 4 (Visits 4 and 7) of each period
Population: FAS. n=18, 18; number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 21 | 22
scores on a scale | -10.67 (21.404) | -7.72 (19.384)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.4999, ANCOVA; Mean Difference (Net) = -4.29, 95% CI 2-sided [-17.13 to 8.54], Standard Error of Mean 6.292

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/30
Other Adverse Events (participants affected / at risk) | 20/28 | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=28) | Placebo (N=30)
Menopause and related conditions (Reproductive system and breast disorders) | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=28) | Placebo (N=30)
Palpitations (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1
Eye pain (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 1
Tongue coated (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Fatigue (General disorders) | 6 | 4
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Eye infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
Disturbance in attention (Nervous system disorders) | 3 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 7 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 2 | 1
Hypnagogic hallucination (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Hot flush (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.